CLINICAL TRIAL: NCT03024918
Title: Unequal Placental Sharing in Monochorionic Diamniotic Twins: an Observational Study to Investigate Prediction and Outcome: the TWINSHARE Study
Brief Title: Unequal Placental Sharing in Monochorionic Diamniotic Twins: an Observational Study
Acronym: TWINSHARE
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S5877
Record Dates: First submitted 2017-01-10; First posted 2017-01-19 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Monochorionic Twins
Keywords: monochorionic; placental sharing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — placental samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MCDA cohort: Unselected monochorionic diamniotic (MCDA) twin pregnancies, included between 11 and 14 weeks of gestation
- TTTS cohort: Pregnancies complicated by twin-twin transfusion syndrome (TTTS) undergoing laser treatment, included at the time of diagnosis or referral
- sIUGR cohort: Pregnancies complicated by selective intrauterine growth restriction (sIUGR), included at the time of diagnosis or referral. We define sIUGR as a discordance in estimated fetal weight of ≥ 20%.

SUMMARY:
This is an observational study in 3 cohorts of monochorionic diamniotic (MCDA) twins. The aim of the study is to assess whether unequal placental sharing can be predicted in pregnancy and whether it is predictive of pregnancy outcome.

DETAILED DESCRIPTION:
In all cohorts, serial ultrasound will be performed during pregnancy. MRI will be offered once during pregnancy. After delivery, placental examination will be performed.

In unselected MCDA twins, the investigators will assess the relationship between unequal placental sharing and the risk of fetal or neonatal loss. The investigators will also establish whether umbilical vein measurements or MRI can be used to predict placental sharing.

In cases complicated by twin-to-twin transfusion syndrome (TTTS), the investigators will look at the association between unequal placental sharing and intrauterine fetal demise after laser surgery.

In cases complicated by selective intra-uterine growth restriction (sIUGR), the the relationship between unequal placental sharing and the risk of fetal or neonatal loss and birth prior to 34 weeks will be assessed.

Furthermore, data on neurological outcome at 2 years of age in all cohorts will be collected.

ELIGIBILITY:
Inclusion Criteria:

* MCDA cohort

  * Ongoing monochorionic diamniotic twin pregnancy between 11 and 14 weeks, as determined by the crown rump length of the larger twin in spontaneous conceptions and by the date of insemination or embryonic age at replacement in pregnancies resulting from subfertility treatment
  * Women aged 18 years or more, who are able to consent
  * Written informed consent to participate in this study, forms being approved by the Ethical Committees
* TTTS cohort

  * Monochorionic diamniotic twin pregnancy, with gestational age defined in the first trimester as mentioned above
  * Complicated by TTTS according to the definition used in the Quintero staging of TTTS (DVP of donor < 2 cm and DVP of receptor > 8 cm before 20 weeks or > 10 cm after 20 weeks
  * Undergoing laser surgery for TTTS
  * Women aged 18 years or more, who are able to consent
  * Written informed consent to participate in this study, forms being approved by the Ethical Committees
* sIUGR cohort

  * Monochorionic diamniotic twin pregnancy, with gestational age defined in the first trimester as mentioned above
  * Complicated by sIUGR defined as a discordance in EFW of ≥ 20%, with the percentage of discordance being calculated as (EFW larger twin - EFW smaller twin)/EFW larger twin x 100.
  * Women aged 18 years or more, who are able to consent
  * Written informed consent to participate in this study, forms being approved by the Ethical Committees

Exclusion Criteria:

* Age < 18 years
* Inability to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population exists of women with a monochorionic twin pregnancy. Three cohorts will be created: a cohort of uncomplicated MCDA twins (included at the first trimester scan), a cohort of MCDA twins complicated by TTTS and undergoing laser surgery (included at the time of diagnosis) and a cohort of MCDA twins complicated by selective growth restriction (included at the time of diagnosis).
Sampling Method: Non-Probability Sample
Enrollment: 393 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MCDA cohort: the association between unequal sharing and risk of fetal or neonatal loss (assessed by review of obstetric and pediatric records) | 2 weeks after expected date of birth
TTTS cohort: the association between unequal sharing and intrauterine fetal death (assessed by review of obstetric records) | 2 weeks after expected date of birth
sIUGR cohort: the association between unequal sharing and risk of fetal or neonatal loss and birth prior to 34 weeks (assessed by review of obstetric and pediatric records) | 2 weeks after expected date of birth

SECONDARY OUTCOMES:
The correlation between prenatal ultrasound and MRI variables and placental sharing as assessed by postnatal imaging (all cohorts) | 2 weeks after expected date of birth
The association between unequal sharing and intact survival (all cohorts) (assessed by review of obstetric and pediatric records and parent questionnaire) | 2 years after expected date of birth

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth Lewi, Study Chair — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lewi L, Jani J, Blickstein I, Huber A, Gucciardo L, Van Mieghem T, Done E, Boes AS, Hecher K, Gratacos E, Lewi P, Deprest J. The outcome of monochorionic diamniotic twin gestations in the era of invasive fetal therapy: a prospective cohort study. Am J Obstet Gynecol. 2008 Nov;199(5):514.e1-8. doi: 10.1016/j.ajog.2008.03.050. Epub 2008 Jun 4. PMID 18533114
- [Background] Lewi L, Gucciardo L, Huber A, Jani J, Van Mieghem T, Done E, Cannie M, Gratacos E, Diemert A, Hecher K, Lewi P, Deprest J. Clinical outcome and placental characteristics of monochorionic diamniotic twin pairs with early- and late-onset discordant growth. Am J Obstet Gynecol. 2008 Nov;199(5):511.e1-7. doi: 10.1016/j.ajog.2008.04.022. Epub 2008 Jun 9. PMID 18539257
- [Background] Cavicchioni O, Yamamoto M, Robyr R, Takahashi Y, Ville Y. Intrauterine fetal demise following laser treatment in twin-to-twin transfusion syndrome. BJOG. 2006 May;113(5):590-4. doi: 10.1111/j.1471-0528.2006.00913.x. Epub 2006 Mar 27. PMID 16579799
- [Background] Lopriore E, Sueters M, Middeldorp JM, Oepkes D, Walther FJ, Vandenbussche FP. Velamentous cord insertion and unequal placental territories in monochorionic twins with and without twin-to-twin-transfusion syndrome. Am J Obstet Gynecol. 2007 Feb;196(2):159.e1-5. doi: 10.1016/j.ajog.2006.10.865. PMID 17306663
- [Background] Lopriore E, Pasman SA, Klumper FJ, Middeldorp JM, Walther FJ, Oepkes D. Placental characteristics in growth-discordant monochorionic twins: a matched case-control study. Placenta. 2012 Mar;33(3):171-4. doi: 10.1016/j.placenta.2011.12.004. Epub 2011 Dec 23. PMID 22197628
- [Background] Aston KI, Peterson CM, Carrell DT. Monozygotic twinning associated with assisted reproductive technologies: a review. Reproduction. 2008 Oct;136(4):377-86. doi: 10.1530/REP-08-0206. Epub 2008 Jun 24. PMID 18577552
- [Background] Lewi L, Deprest J, Hecher K. The vascular anastomoses in monochorionic twin pregnancies and their clinical consequences. Am J Obstet Gynecol. 2013 Jan;208(1):19-30. doi: 10.1016/j.ajog.2012.09.025. Epub 2012 Sep 28. PMID 23103301
- [Background] Kent EM, Breathnach FM, Gillan JE, McAuliffe FM, Geary MP, Daly S, Higgins JR, Dornan J, Morrison JJ, Burke G, Higgins S, Carroll S, Dicker P, Manning F, Malone FD. Placental cord insertion and birthweight discordance in twin pregnancies: results of the national prospective ESPRiT Study. Am J Obstet Gynecol. 2011 Oct;205(4):376.e1-7. doi: 10.1016/j.ajog.2011.06.077. Epub 2011 Jun 25. PMID 21864823
- [Background] Monk D. Genomic imprinting in the human placenta. Am J Obstet Gynecol. 2015 Oct;213(4 Suppl):S152-62. doi: 10.1016/j.ajog.2015.06.032. PMID 26428495
- [Background] Su EJ. Role of the fetoplacental endothelium in fetal growth restriction with abnormal umbilical artery Doppler velocimetry. Am J Obstet Gynecol. 2015 Oct;213(4 Suppl):S123-30. doi: 10.1016/j.ajog.2015.06.038. PMID 26428491
- [Background] Su EJ, Xin H, Yin P, Dyson M, Coon J, Farrow KN, Mestan KK, Ernst LM. Impaired fetoplacental angiogenesis in growth-restricted fetuses with abnormal umbilical artery doppler velocimetry is mediated by aryl hydrocarbon receptor nuclear translocator (ARNT). J Clin Endocrinol Metab. 2015 Jan;100(1):E30-40. doi: 10.1210/jc.2014-2385. PMID 25343232
- [Background] Gratacos E, Lewi L, Munoz B, Acosta-Rojas R, Hernandez-Andrade E, Martinez JM, Carreras E, Deprest J. A classification system for selective intrauterine growth restriction in monochorionic pregnancies according to umbilical artery Doppler flow in the smaller twin. Ultrasound Obstet Gynecol. 2007 Jul;30(1):28-34. doi: 10.1002/uog.4046. PMID 17542039
- [Background] Ishii K, Murakoshi T, Takahashi Y, Shinno T, Matsushita M, Naruse H, Torii Y, Sumie M, Nakata M. Perinatal outcome of monochorionic twins with selective intrauterine growth restriction and different types of umbilical artery Doppler under expectant management. Fetal Diagn Ther. 2009;26(3):157-61. doi: 10.1159/000253880. Epub 2009 Oct 28. PMID 19864880
- [Background] Gratacos E, Carreras E, Becker J, Lewi L, Enriquez G, Perapoch J, Higueras T, Cabero L, Deprest J. Prevalence of neurological damage in monochorionic twins with selective intrauterine growth restriction and intermittent absent or reversed end-diastolic umbilical artery flow. Ultrasound Obstet Gynecol. 2004 Aug;24(2):159-63. doi: 10.1002/uog.1105. PMID 15287053
- [Background] Peeva G, Bower S, Orosz L, Chaveeva P, Akolekar R, Nicolaides KH. Endoscopic Placental Laser Coagulation in Monochorionic Diamniotic Twins with Type II Selective Fetal Growth Restriction. Fetal Diagn Ther. 2015;38(2):86-93. doi: 10.1159/000374109. Epub 2015 Apr 15. PMID 25896405
- [Background] Parra-Cordero M, Bennasar M, Martinez JM, Eixarch E, Torres X, Gratacos E. Cord Occlusion in Monochorionic Twins with Early Selective Intrauterine Growth Restriction and Abnormal Umbilical Artery Doppler: A Consecutive Series of 90 Cases. Fetal Diagn Ther. 2016;39(3):186-91. doi: 10.1159/000439023. Epub 2015 Sep 8. PMID 26344150
- [Background] Chalouhi GE, Marangoni MA, Quibel T, Deloison B, Benzina N, Essaoui M, Al Ibrahim A, Stirnemann JJ, Salomon LJ, Ville Y. Active management of selective intrauterine growth restriction with abnormal Doppler in monochorionic diamniotic twin pregnancies diagnosed in the second trimester of pregnancy. Prenat Diagn. 2013 Feb;33(2):109-15. doi: 10.1002/pd.4031. Epub 2012 Dec 26. PMID 23280487
- [Background] Bonel HM, Stolz B, Diedrichsen L, Frei K, Saar B, Tutschek B, Raio L, Surbek D, Srivastav S, Nelle M, Slotboom J, Wiest R. Diffusion-weighted MR imaging of the placenta in fetuses with placental insufficiency. Radiology. 2010 Dec;257(3):810-9. doi: 10.1148/radiol.10092283. PMID 21084415
- [Background] Derwig I, Lythgoe DJ, Barker GJ, Poon L, Gowland P, Yeung R, Zelaya F, Nicolaides K. Association of placental perfusion, as assessed by magnetic resonance imaging and uterine artery Doppler ultrasound, and its relationship to pregnancy outcome. Placenta. 2013 Oct;34(10):885-91. doi: 10.1016/j.placenta.2013.07.006. Epub 2013 Aug 9. PMID 23937958
- [Background] Lewi L, Cannie M, Blickstein I, Jani J, Huber A, Hecher K, Dymarkowski S, Gratacos E, Lewi P, Deprest J. Placental sharing, birthweight discordance, and vascular anastomoses in monochorionic diamniotic twin placentas. Am J Obstet Gynecol. 2007 Dec;197(6):587.e1-8. doi: 10.1016/j.ajog.2007.05.009. PMID 18060944
- [Background] De Paepe ME, Shapiro S, Young L, Luks FI. Placental characteristics of selective birth weight discordance in diamniotic-monochorionic twin gestations. Placenta. 2010 May;31(5):380-6. doi: 10.1016/j.placenta.2010.02.018. Epub 2010 Mar 19. PMID 20303588
- [Background] Janzen C, Lei MY, Cho J, Sullivan P, Shin BC, Devaskar SU. Placental glucose transporter 3 (GLUT3) is up-regulated in human pregnancies complicated by late-onset intrauterine growth restriction. Placenta. 2013 Nov;34(11):1072-8. doi: 10.1016/j.placenta.2013.08.010. Epub 2013 Aug 28. PMID 24011442
- [Background] Yung HW, Calabrese S, Hynx D, Hemmings BA, Cetin I, Charnock-Jones DS, Burton GJ. Evidence of placental translation inhibition and endoplasmic reticulum stress in the etiology of human intrauterine growth restriction. Am J Pathol. 2008 Aug;173(2):451-62. doi: 10.2353/ajpath.2008.071193. Epub 2008 Jun 26. PMID 18583310
- [Background] Kent EM, Breathnach FM, Gillan JE, McAuliffe FM, Geary MP, Daly S, Higgins JR, Hunter A, Morrison JJ, Burke G, Higgins S, Carroll S, Dicker P, Manning F, Tully E, Malone FD. Placental pathology, birthweight discordance, and growth restriction in twin pregnancy: results of the ESPRiT Study. Am J Obstet Gynecol. 2012 Sep;207(3):220.e1-5. doi: 10.1016/j.ajog.2012.06.022. Epub 2012 Jul 25. PMID 22835491
- [Background] Zhang GL, He ZM, Shi XM, Gou CY, Gao Y, Fang Q. Discordant HIF1A mRNA levels and oxidative stress in placental shares of monochorionic twins with selective intra-uterine growth restriction. Placenta. 2015 Mar;36(3):297-303. doi: 10.1016/j.placenta.2014.12.019. Epub 2014 Dec 30. PMID 25573093
- [Background] Schrey S, Kingdom J, Baczyk D, Fitzgerald B, Keating S, Ryan G, Drewlo S. Leptin is differentially expressed and epigenetically regulated across monochorionic twin placenta with discordant fetal growth. Mol Hum Reprod. 2013 Nov;19(11):764-72. doi: 10.1093/molehr/gat048. Epub 2013 Jul 4. PMID 23832168
- [Background] Salomon LJ, Alfirevic Z, Bilardo CM, Chalouhi GE, Ghi T, Kagan KO, Lau TK, Papageorghiou AT, Raine-Fenning NJ, Stirnemann J, Suresh S, Tabor A, Timor-Tritsch IE, Toi A, Yeo G. ISUOG practice guidelines: performance of first-trimester fetal ultrasound scan. Ultrasound Obstet Gynecol. 2013 Jan;41(1):102-13. doi: 10.1002/uog.12342. No abstract available. PMID 23280739
- [Background] Salomon LJ, Alfirevic Z, Berghella V, Bilardo C, Hernandez-Andrade E, Johnsen SL, Kalache K, Leung KY, Malinger G, Munoz H, Prefumo F, Toi A, Lee W; ISUOG Clinical Standards Committee. Practice guidelines for performance of the routine mid-trimester fetal ultrasound scan. Ultrasound Obstet Gynecol. 2011 Jan;37(1):116-26. doi: 10.1002/uog.8831. No abstract available. PMID 20842655
- [Background] Liao TB, Nomura RM, Liao AW, Francisco RP, Zugaib M. Fetal venous circulation in monochorionic twin pregnancies with placental insufficiency: prediction of acidemia at birth or intrauterine fetal death. Ultrasound Obstet Gynecol. 2014 Apr;43(4):426-31. doi: 10.1002/uog.12549. Epub 2014 Mar 12. PMID 23828752
- [Background] Levine D, Zuo C, Faro CB, Chen Q. Potential heating effect in the gravid uterus during MR HASTE imaging. J Magn Reson Imaging. 2001 Jun;13(6):856-61. doi: 10.1002/jmri.1122. PMID 11382944
- [Background] Strizek B, Jani JC, Mucyo E, De Keyzer F, Pauwels I, Ziane S, Mansbach AL, Deltenre P, Cos T, Cannie MM. Safety of MR Imaging at 1.5 T in Fetuses: A Retrospective Case-Control Study of Birth Weights and the Effects of Acoustic Noise. Radiology. 2015 May;275(2):530-7. doi: 10.1148/radiol.14141382. Epub 2015 Jan 7. PMID 25575119
- See also: Study website — http://www.monochorionictwins.org